CLINICAL TRIAL: NCT07285629
Title: Evaluating the Safety and Efficacy of Injectable Combination Klotho and Follistatin Plasmid Gene Therapy in Humans -- An Interventional, Non-Placebo Controlled Pilot Phase Study
Brief Title: Safety and Efficacy of Klotho and Follistatin Gene Therapy
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Minicircle (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GIFIRB202507313
Record Dates: First submitted 2025-11-27; First posted 2025-12-16 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Healthy Adults
Keywords: klotho; follistatin; nonviral; gene therapy; plasmid
MeSH Terms: interventions — Follistatin

STUDY DESIGN:
Intervention Model Description: Non-placebo-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention with Cognitive/Health battery before and after (Experimental): This arm includes cognitive and health battery pre- and post-intervention of the gene therapy
  Interventions: Genetic: Follistatin and klotho gene therapy

INTERVENTIONS:
Genetic: Follistatin and klotho gene therapy — Injection of nonviral plasmid-delivered follistatin and klotho gene therapy

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of a combination klotho and follistatin gene therapy, delivered via a nonviral plasmid in healthy adult volunteers. Additionally, this study seeks to understand the cognitive and health benefits of this gene therapy.

DETAILED DESCRIPTION:
Healthy participants will take part in cognitive and health testing before and after administration of plasmid-delivered nonviral klotho and follistatin gene therapy. The method of administration will be subcutaneous injection into abdominal fat deposits. Klotho and follistatin plasmid gene therapy have the potential to improve physical function, cognitive function, kidney function, body composition, epigenetic age, and subjective well being.

Note that the investigational product will be administered at a site outside of the U.S. which is not under FDA jurisdiction, and only non-treatment pre/post outcome assessments (e.g., cognitive assessments or blood sample collection) occur at the U.S. site.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 50 to 80 years
* General good health
* Willing to comply with all study-related procedures and visits
* Participant is open to morphological change
* If female, participant agrees to maintain contraception
* If female, participant agrees to take a pregnancy test
* If female, participant agrees to a pregnancy waiver

Exclusion Criteria:

* Currently enrolled in another clinical trial
* History of cancer, autoimmune disease, or chronic kidney/liver disease
* Use of immunosuppressive therapy
* Pregnant or breastfeeding
* Women of childbearing potential who are unwilling or unable to use effective contraception for the duration of the study.
* Regular use of NMDA (N-methyl-D-aspartate) antagonists (i.e., memantine, ketamine, etc.)
* Regular use of antiplatelet medications (i.e., aspirin)
* Any medical or psychiatric condition that could interfere with participation or pose safety concerns
* Unwilling or unable to provide informed consent

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Concentration of Serum α-Klotho Measured by Enzyme-Linked Immunosorbent Assay (ELISA) (pg/mL) | From 1 month prior to treatment to 3 months after treatment (5 timepoints)
  Serum α-Klotho protein concentration will be quantified using a validated ELISA. Results will be determined from picograms per milliliter (pg/mL) for each participant at each time point. Higher or lower values have no inherent directionality and will be interpreted in study context.
Concentration of Serum Follistatin Measured by Enzyme-Linked Immunosorbent Assay (ELISA) (pg/mL) | From 1 month prior to treatment to 3 months after treatment (5 timepoints)
  Serum follistatin concentration will be quantified using a validated ELISA. Results will be reported as picograms per milliliter (pg/mL) for each participant at each time point. Higher or lower values have no inherent directionality and will be interpreted in study context.
Number and Percentage of Participants Experiencing Treatment-Emergent Adverse Events as Assessed by Patient-Reported Outcomes Version of Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Within 1 week after treatment and then 1 month, 2 months, and 3 months after treatment
  Assessed through a checklist version of the PRO-CTCAE with each symptom options being none, mild, moderate, or severe. Items will be scored with 0, 1, 2, 3 respectively. Item responses will be summarized as number and percentage of participants experiencing each adverse event by system/organ class. High scores indicate highest severity of symptoms and low scores indicate no symptoms.

SECONDARY OUTCOMES:
Change From Baseline in World Health Organization Quality of Life Brief Version (WHOQOL-BREF) Domain Scores (0-100) | From 1 month prior to treatment to 3 months after treatment (5 timepoints)
  The WHOQOL-BREF is a self-report questionnaire that includes four domains: Physical Health, Psychological, Social Relationships, and Environment. Each domain score is transformed to a 0-100 scale, with higher scores indicating better quality of life. Changes from baseline will be examined per domain.
Change From Baseline in Pattern Comparison Processing Speed Test T-Score (Mean 50 ± 10) | From 1 month prior to treatment to 3 months after treatment (4 timepoints)
  The Pattern Comparison Processing Speed Test measures processing speed using age-adjusted T-scores (mean 50, SD 10). Higher scores reflect faster cognitive processing. Changes from baseline will be analyzed per participant and time point.
Change From Baseline in Picture Sequence Memory Test T-Score, Forms A and B (Mean 50 ± 10) | From 1 month prior to treatment to 3 months after treatment (4 timepoints)
  Picture Sequence Memory Test evaluates episodic memory. Each form (A and B) yields an age-adjusted T-score (mean 50, SD 10). Higher scores indicate better memory performance. Forms A and B will be averaged.
Change From Baseline in Flanker Inhibitory Control and Attention Test T-Score (Mean 50 ± 10) | From 1 month prior to treatment to 3 months after treatment (4 timepoints)
  The Flanker Inhibitory Control and Attention Test measures inhibitory control and attention. Scores are age-adjusted T-scores (mean 50, SD 10). Higher scores indicate better performance. Changes from baseline will be analyzed per participant and time point.
Change From Baseline in Dimensional Change Card Sort Test T-Score (Mean 50 ± 10) | From 1 month prior to treatment to 3 months after treatment (4 timepoints)
  The Dimensional Change Card Sort Test assesses cognitive flexibility. Scores are age-adjusted T-scores (mean 50, SD 10). Higher scores indicate better executive function. Changes from baseline will be analyzed per participant and time point.
Change From Baseline in Picture Vocabulary Test T-Score (Mean 50 ± 10) | From 1 month prior to treatment to 3 months after treatment (5 timepoints)
  Picture Vocabulary Test measures receptive vocabulary. Results are expressed as age-adjusted T-scores (mean 50, SD 10), with higher scores indicating better performance. Change from baseline will be analyzed per participant and time point.
Epigenetic Biological Age Estimated From Whole-Genome Deoxyribonucleic Acid (DNA) Methylation Profiles (change from baseline) (years) | From 1 month prior to treatment to 3 months after treatment (5 timepoints)
  Whole-blood DNA methylation will be measured using bisulfite sequencing performed by Generation Lab. Epigenetic biological age will be computed from these methylation data using validated algorithms. Age estimates will be expressed in years. Lower epigenetic age relative to chronological age indicates younger biological status.
Timed one leg stance change from baseline (seconds) | From 1 month prior to treatment to 3 months after treatment (4 timepoints)
  Duration (seconds) that the participant can maintain an unsupported one-leg stance on the left and right leg separately, measured from the point of foot lift until loss of balance or foot contact with the ground.
Change from baseline in number of squats performed (count) | From 1 month prior to treatment to 3 months after treatment (4 timepoints)
  Total number of full squats the participant can complete with proper form within a continuous, unassisted trial, measured from the start of movement until the participant stops or is unable to continue.
Change from baseline in number of push-ups performed (count) | From 1 month prior to treatment to 3 months after treatment (4 timepoints)
  Total number of standard push-ups completed with proper form in a continuous trial, counted from the first repetition until the participant stops or is unable to continue.
Number of sit-ups performed (change from baseline) (count) | From 1 month prior to treatment to 3 months after treatment (4 timepoints)
  Total number of sit-ups the participant can complete with proper form in a continuous trial, measured from the first repetition until the participant stops or is unable to continue.
Change from Baseline: Concentration of High-Sensitivity C-Reactive Protein (hs-CRP) Measured by Immunoturbidimetric Assay (mg/L) | From 1 month prior to treatment to 3 months after treatment (5 timepoints)
  hs-CRP will be measured using an immunoturbidimetric assay and expressed in mg/L. hs-CRP is a marker of systemic inflammation and cardiovascular risk.
Concentration of Ionized Calcium Measured by Ion-Selective Electrode (mmol/L) | From 1 month prior to treatment to 3 months after treatment (5 timepoints)
  Ionized calcium will be measured using an ion-selective electrode analyzer. Results will be reported in millimoles per liter (mmol/L) and represent physiologically active calcium fraction.
Concentration of Serum Cystatin C Measured by Immunoassay (mg/L) | From 1 month prior to treatment to 3 months after treatment (5 timepoints)
  Serum Cystatin C will be measured using a standardized immunoassay and reported in mg/L for each participant and time point. Cystatin C is a biomarker of glomerular filtration rate and provides a mechanistic link between α-Klotho activity and renal function.
Concentration of Serum Phosphorus Measured by Clinical Chemistry Analyzer (mg/dL) | From 1 month prior to treatment to 3 months after treatment (5 timepoints)
  Serum inorganic phosphorus will be measured on a standard clinical chemistry analyzer. Results will be reported in mg/dL for each participant and time point. Phosphorus levels reflect systemic phosphate homeostasis influenced by α-Klotho and FGF23 activity.
Urinary Phosphate Excretion Measured by Clinical Chemistry Assay (mg/24 h or mg/g Creatinine) | From 1 month prior to treatment to 3 months after treatment (5 timepoints)
  Urinary phosphate will be assessed using a validated chemistry assay. Will be expressed either as total phosphate excretion in milligrams per 24 hours (mg/24 h) or as the phosphate-to-creatinine ratio (mg phosphate per g creatinine). This measure reflects renal handling of phosphate and functional effects of α-Klotho on phosphate excretion.
Concentration of Intact Parathyroid Hormone Measured by Two-Site Immunoassay (pg/mL) | From 1 month prior to treatment to 3 months after treatment (5 timepoints)
  Intact Parathyroid Hormone (PTH) will be measured in serum using a two-site immunoassay that detects the full-length molecule. Results will be reported in picograms per milliliter (pg/mL) per participant and time point. PTH reflects parathyroid activity within the α-Klotho-FGF23-vitamin D feedback pathway.
Concentration of Serum 1,25-Dihydroxyvitamin D (Calcitriol) Measured by Liquid Chromatography-Tandem Mass Spectrometry (pg/mL) | From 1 month prior to treatment to 3 months after treatment (5 timepoints)
  Serum 1,25-dihydroxyvitamin D (calcitriol) will be quantified using liquid chromatography-tandem mass spectrometry (LC-MS/MS). Concentrations will be expressed in picograms per milliliter (pg/mL). This hormone regulates calcium and phosphate balance and is a downstream marker of α-Klotho-FGF23-PTH axis modulation.
Comprehensive Metabolic Panel (Safety Laboratory Assessment) | From 1 month prior to treatment to 3 months after treatment (5 timepoints)
  A standard comprehensive metabolic panel (CMP) will be collected to evaluate general metabolic and organ function for safety monitoring. The standard panel includes 14 markers: Glucose, calcium, sodium, potassium, chloride, bicarbonate, blood urea nitrogen, creatinine (serum), albumin, total protein, alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase, and total bilirubin. Individual components will be assessed clinically to ensure no major changes to health stability but these will not analyzed as specific study endpoints.
Concentration of Platelet Factor 4 (PF4) Measured by Enzyme-Linked Immunosorbent Assay (ELISA) (ng/mL or OD Units) | From 1 month prior to treatment to 3 months after treatment (5 timepoints)
  Platelet Factor 4 (PF4) will be measured using a validated ELISA and reported as nanograms per milliliter (ng/mL) or optical density (OD) units. PF4 is a marker of platelet activation and potential immune-mediated coagulation effects.
Cardio IQ® Fibrinogen Antigen (mg/dL) | From 1 month prior to treatment to 3 months after treatment (5 timepoints)
  Fibrinogen antigen concentration will be measured by nephelometry using the Cardio IQ® assay. Reported in milligrams per deciliter (mg/dL).
Hemoglobin A1c (%) change from baseline | From 1 month prior to treatment to 3 months after treatment (5 timepoints)
  Hemoglobin A1c (HbA1c) will be measured by standardized assay methods and reported as percent (%). Estimated average glucose (eAG) will be reported alongside HbA1c for interpretability only and will be derived from the HbA1c value using a validated conversion formula. eAG is not independently measured. Change from baseline HbA1c will be reported as a percentage and the corresponding eAG value will be included for interpretability.
Homocysteine change from baseline (µmol/L) | From 1 month prior to treatment to 3 months after treatment (5 timepoints)
  Plasma homocysteine concentration will be measured by immunoassay or chromatography-based methods and reported in micromoles per liter (µmol/L).
Asymmetric and Symmetric Dimethylarginine (ADMA/SDMA) change from baseline (µmol/L) | From 1 month prior to treatment to 3 months after treatment (5 timepoints)
  Plasma ADMA and SDMA will be quantified by mass spectrometry-based assay and reported in micromoles per liter (µmol/L).
Serum Interleukin-6 (IL-6) change from baseline (pg/mL) | From 1 month prior to treatment to 3 months after treatment (5 timepoints)
  Serum IL-6 levels will be measured by high-sensitivity immunoassay and reported in picograms per milliliter (pg/mL).
Tumor Necrosis Factor-α (TNF-α) change from baseline (pg/mL) | From 1 month prior to treatment to 3 months after treatment (5 timepoints)
  Serum TNF-α concentration will be measured by immunoassay and reported in picograms per milliliter (pg/mL).
Serum Interleukin-1β (IL-1β) change from baseline (pg/mL) | From 1 month prior to treatment to 3 months after treatment (5 timepoints)
  Serum IL-1β levels will be quantified using a cytokine immunoassay and reported in picograms per milliliter (pg/mL).
Serum Interferon-γ (IFN-γ) (pg/mL) | From 1 month prior to treatment to 3 months after treatment (5 timepoints)
  Plasma IFN-γ concentration will be measured using an immunoassay and reported in picograms per milliliter (pg/mL).
Serum Interleukin-10 (IL-10) (pg/mL) | From 1 month prior to treatment to 3 months after treatment (5 timepoints)
  Serum IL-10 levels will be measured by cytokine immunoassay and reported in picograms per milliliter (pg/mL).
Myostatin (ng/mL) | From 1 month prior to treatment to 3 months after treatment (5 timepoints)
  Serum myostatin concentration will be measured using a validated immunoassay and reported in nanograms per milliliter (ng/mL).
Activin A (pg/mL) | From 1 month prior to treatment to 3 months after treatment (5 timepoints)
  Serum activin A will be quantified by immunoassay and reported in picograms per milliliter (pg/mL).
Insulin-Like Growth Factor-1 (IGF-1) (ng/mL) | From 1 month prior to treatment to 3 months after treatment (5 timepoints)
  Serum IGF-1 will be measured using a standardized immunoassay with age-adjusted calibration and reported in nanograms per milliliter (ng/mL).

CONTACTS AND LOCATIONS:
Locations (2):
- Apeiron Center, Austin, Texas, United States
- Global Alliance of Regenerative Medicine (GARM) Clinic, Roatán, Bay Islands, Honduras

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be made available along with a data dictionary describing each variable. If the study results in multiple publications, the IPD corresponding to the measures reported in each publication will be shared upon that publication. The complete trial dataset, if anything is remaining, will be made available once all results have been published. Supporting documentation shared will include study protocol, statistical analysis plan, informed consent forms, and analytic code.
Time Frame: Data will be made available upon publication and will be available indefinitely.
Access Criteria: Data will be made available to anyone who wishes to access it in an online repository at Zenodo (https://zenodo.org/). The types of data shared will include de-identified data of pre- and post-treatment values for the following measures: serum Klotho levels; serum Follistatin levels; kidney and blood safety panels; questionnaires and adverse event reporting data (all check box questions; however, any open-ended answer data will reviewed to ensure they cannot be used to identify an individual participant - final judgments will be made by the study central coordinator); quantitative muscle function outcomes; all NIH-toolbox measures; epigenetic age.